CLINICAL TRIAL: NCT06410391
Title: Fetal Brain Sonographic Measurements and Normograms in Healthy Fetuses During Second and Third Trimesters
Brief Title: Fetal Brain Ultrasound
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal M.fekry, Lecturer of Obs& Gyn. Specialist of Urogynecology, Assiut University
Other Study IDs: FBUS
Record Dates: First submitted 2024-05-03; First posted 2024-05-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-06

CONDITIONS: Fetal Anomaly
MeSH Terms: conditions — Congenital Abnormalities | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: Ultrasound — Gestational age, biparietal diameter and head circumference are measured. then 2 techniques are used according to the 2007 International Society of Ultrasound in Obstetrics and Gynecology guidelines for a US evaluation of the fetal central nervous system (CNS) (10) : 1- the axial transventricular technique including the posterior portions of the lateral ventricles, falx, CSP, and Frontal horn 2- the trans-cerebellar technique, including the cerebellum, cisternal magna, cerebellar peduncles, CSP, and FHs. CSP visualization and width, FH width, anterior horn width (AHW), center from the horn distance (CFHD), upside and downside measurement.
  The corpus callosum is identified in the midsagittal plane. The image selected for CC measurement in addition to cerebellar vermis and cisterna magna

SUMMARY:
The aim of our study is to determine the range of frontal horn sizes (both upside and downside) in healthy fetuses over gestation and to determine how far FHs are from the midline . Also to determine the range of cavum septi pellucidi and Corpus callosum sizes . Also, to determine whether the maternal body mass index (BMI) affects rates of visualized and non-visualized CSP and CC.

DETAILED DESCRIPTION:
Fetal central nervous system (CNS) abnormalities are among the most commonly encountered congenital abnormalities . Many different methods can be used to obtain prenatal diagnoses, including ultrasound (US), which is one of the most commonly used methods .Neonatal survival rates have increased over the last decades leading to increased number of infants with adverse neurodevelopmental outcomes, including cognitive, motor impairments and behavioral and learning difficulties later in life . Recent studies demonstrated that signs of abnormal neurological development are already present at birth .

Frontal horns (FHs) are the most anterior portions of the lateral ventricles, on each side the cavum septi pellucidi (CSP). In accordance with practice parameters released as early as 1985 by the American Institute of Ultrasound in Medicine, American College of Obstetrics and Gynecology, and Society of Radiologists in Ultrasound, the CSP is examined in screening fetal ultrasound (US) examinations in the biparietal diameter view . Frontal horns (FH) are also visualized in the same plane. Abnormal morphologic characteristics of the FHs such as enlargement, squaring, spearing, and splaying may have an association with congenital intracranial anomalies such as holoprosencephaly, schizencephaly and agenesis of the corpus callosum .

The corpus callosum (CC) is the largest interhemispheric white matter commissure of the human brain . It is a sensitive indicator of normal brain development and maturation

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman 15 weeks to 36 weeks

Exclusion Criteria:

* congenital malformations
* Multiple pregnancy
* intrauterine infection
* fetuses with Fetal growth restriction

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All healthy pregnant women came to fetal medicine unit at 15 to 36 weeks
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Determine the range of lateral ventricles diameter in healthy fetuses at different gestational ages., | 5 months
  Diameter of Lateral ventricles measured by ultrasound in millimeters

SECONDARY OUTCOMES:
measurement of Cavum septum and Corpus callosum | 5 months
  Length of Cavum septum and Corpus callosum measured by ultrasound in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No